CLINICAL TRIAL: NCT00721604
Title: Prediction of Volume Expansion Effectiveness in Hypotensive Critically Ill Patients.
Brief Title: Fluid Responsiveness Prediction at the Bedside
Status: Completed | Type: Observational
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Natalini Giuseppe, FPoliambulanza
Other Study IDs: FP-TIP-03
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Hypotension; Shock
Keywords: shock; fluid responsiveness; volume expansion
MeSH Terms: conditions — Hypotension; Shock | interventions — Hypodermoclysis; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with mean arterial pressure lower than 65 mmHg
  Interventions: Drug: fluid administration

INTERVENTIONS:
Drug: fluid administration — two consecutive infusions of 6% hydroxyethyl starch at the dosage 7 ml/kg over 30 minutes (total 14 ml/kg in 60 minutes)
  Other Names: Haes Steril, Fresenius Kabi

SUMMARY:
The purpose of this study is to verify the accuracy and applicability of predictors of fluid administration efficacy in hypotensive critically ill patients.

DETAILED DESCRIPTION:
Severe hypotension is a common life-threatening conditions in critically ill patients. Discriminating between the need for volume expansion or inotropic/vasoactive support is a main clinical goal. Pulse pressure variation are an accurate index of fluid responsiveness, but it needs controlled mechanical ventilation with a tidal volume of at least 8 ml/kg and absence of arrhythmias. This could limit its clinical applicability. Moreover pulse pressure variation accurately predicted cardiac output increment. However the cardiac output increase is not a clinically relevant target in absence of low cardiac output.

The objectives of the present protocol are: 1) to calculate the accuracy of cardiovascular and renal variables to predict either arterial pressure increase or clinically relevant improvement after fluid administration and 2) to verify how often dynamic indices could be applied in clinical practice.

Arterial pressure increase is defined by mean arterial pressure above 65 mmHg or an increment greater than 20 % respect to basal value. Clinically relevant improvement is defined by restoring adequate values of arterial pressure or cardiac index or diuresis or central venous saturation if they are inadequate before fluid administration. These adequate values are 65 mmHg for mean arterial pressure, 2.5 l.min-1.m-2 for cardiac index, 0.5 ml.kg-1.h-1 for the diuresis, 70 % for central venous saturation.

ELIGIBILITY:
Inclusion Criteria:

* mean arterial pressure lower than 65 mmHg

Exclusion Criteria:

* fluid overload
* mean arterial pressure lower than 45 mmHg and mandatory immediate treatment
* active bleeding
* hemoglobin lower than 8 g.dl-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypotensive patients in a General Intensive Care Unit of a University-affiliated hospital. Patients can be recruited only if they have both arterial and central venous catheters
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
area under ROC curve of pulse pressure variation before volume expansion and their positive and negative predictive values; responders are patients increasing mean arterial pressure | one hour after the end of fluid administration

SECONDARY OUTCOMES:
area under ROC curve of pulse plethysmographic variation before volume expansion and their positive and negative predictive values; responders are patients increasing mean arterial pressure | one hour after the end of fluid administration
area under ROC curve of pulse pressure variation before volume expansion, positive and negative predictive values; responders are patients showing any clinical improvement | one hour after the end of fluid administration
area under ROC curve of pulse plethysmographic variation before volume expansion, positive and negative predictive values; responders are patients showing any clinical improvement | one hour after the end of fluid administration
area under ROC curve of central venous pressure before volume expansion and their positive and negative predictive values; responders are patients increasing mean arterial pressure | one hour after the end of fluid administration
area under ROC curve of central venous pressure before volume expansion, positive and negative predictive values; responders are patients showing any clinical improvement | one hour after the end of fluid administration
area under ROC curve of central venous saturation before volume expansion, positive and negative predictive values; responders are patients showing any clinical improvement | one hour after the end of fluid administration
area under ROC curve of central-arterial PCO2 pressure difference before volume expansion, positive and negative predictive values; responders are patients showing any clinical improvement | one hour after the end of fluid administration
area under ROC curve of arterial lactate before volume expansion, positive and negative predictive values; responders are patients showing any clinical improvement | one hour after the end of fluid administration
area under ROC curve of fractional excretion of sodium before volume expansion, positive and negative predictive values; responders are patients showing any clinical improvement | one hour after the end of fluid administration
area under ROC curve of sodium/potassium urinary ratio before volume expansion, positive and negative predictive values; responders are patients showing any clinical improvement | one hour after the end of fluid administration
comparison between the number of patients with criteria for pulse pressure variation calculation and the number of patients with other predictive variables | one hour after the end of fluid administration
estimation of variables independently associated to arterial pressure increase | one hour after the end of fluid administration
estimation of variables independently associated to clinically relevant improvement | one hour after the end of fluid administration

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Natalini, MD, Principal Investigator — Fondazione Poliambulanza Istituto Ospedaliero
Locations (1):
- Intensive Care Unit, Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Italy

REFERENCES:
- [Derived] Natalini G, Rosano A, Militano CR, Di Maio A, Ferretti P, Bertelli M, de Giuli F, Bernardini A. Prediction of arterial pressure increase after fluid challenge. BMC Anesthesiol. 2012 Mar 5;12:3. doi: 10.1186/1471-2253-12-3. PMID 22390818